CLINICAL TRIAL: NCT04977804
Title: Effects of Blood Flow Restriction During Multiple-joint Eccentric Resistance Training on Muscle Morphology and Function of the Lower Body.
Brief Title: Eccentric Resistance Training With Blood Flow Restriction on Muscle Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: A key faculty at our college who was helping with the project left the college.
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Brennan Thompson, Principal Investigator, Utah State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12042b
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Blood Flow Restriction
Keywords: resistance training; muscle function; quadriceps; eccentric strength; vertical jump; muscle quality; muscle hypertrophy; eccentric training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two group, randomized parallel group design.
Who Masked: Outcomes Assessor
Masking Description: The person assessing the outcome measures will be blinded to the group designation of the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric only training (Active Comparator): This is the experimental control; where this group will be used as the standard active comparison condition.
  Interventions: Other: Exercise
- Eccentric plus blood-flow restriction (Experimental): This is the experimental condition involving the eccentric resistance training with blood flow restriction.
  Interventions: Other: Eccentric plus blood-flow restriction

INTERVENTIONS:
Other: Exercise — The interventions are a form or exercise, specifically resistance exercise.
  Arms: Eccentric only training
Other: Eccentric plus blood-flow restriction — Eccentric plus blood-flow restriction
  Arms: Eccentric plus blood-flow restriction

SUMMARY:
The study will determine the effects of adding blood flow restriction to eccentric training to assess whether this increases the improvements of muscle strength and size.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to two groups: an eccentric only resistance training group or an eccentric training plus blood flow restriction group. Subjects will train at a moderately low intensity on a multiple-joint eccentric device. Those in the blood flow restriction will wear blood flow restriction cuffs on their upper thighs to reduce blood flow during the brief protocol. The training session will occur twice per week and will last ~5 minutes, including a one minute warm up, a one minute cool down and a three minute workout phase. The training program will last 7 weeks. Testing will be conducted at baseline (following a one session familiarization), 4 weeks and after the end of the 7 week training period. Assessments will focus on muscle strength, function, and morphology (size).

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* currently engaged in some form of resistance training between 1-3 times per week
* must have been training aerobically, but no more than 3 hours a week for the past six months

Exclusion Criteria:

* Must not have had any surgery of the lower limbs within the past 1 year period
* Must not have any neuromuscular disorder (e.g., Muscular dystrophy etc.)
* < 76 inches tall (in order to fit on the training machine)
* Maximal strength of < 725 lbs for the eccentric training device
* If any of the subjects are pregnant or plan to be pregnant in the duration of the protocol.

For those randomized to the BFR group, if any of the subject's thighs are too large for the BFR cuffs (greater than 68 cm).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Eccentron maximal muscle strength | 7 weeks
  Eccentric muscle strength will be assessed via Eccentron (BTE Technologies, Inc., USA), an seated isokinetic dynamometer.
Local muscle hypertrophy | 7 weeks
  Muscle size changes of the quadriceps muscle measured an ultrasound device (GE NextGen LOGIQ, Tampa, Florida, USA).
Muscle mass | 7 weeks
  dual energy x-ray absorptiometry device (DEXA) the Hologic Horizon W Dual X-ray absorptiometry (Hologic Canada ULC, Mississauga, ON, Canada) will be used to assess appendicular (lower body) mean mass.
Muscle function | 7 weeks
  Vertical jump height will assess 3 maximal countermovement attempts on a jump mat (Just Jump Technologies, Huntsville, AL, USA) that measures jump height based on flight time.

SECONDARY OUTCOMES:
Muscle soreness | 7 weeks
  local muscle soreness will be assessed throughout the duration of the intervention period using a Wagner force algometer.

CONTACTS AND LOCATIONS:
Overall Officials: Brennan J Thompson, PhD, Principal Investigator — Utah State Univeristy
Locations (1):
- Utah State Universtiy, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No